CLINICAL TRIAL: NCT00192855
Title: Entacapone Augmentation for Schizophrenia- A Randomized Controlled Trial
Brief Title: Entacapone Augmentation for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Ehud Klein, MD, Head Department of Psychiatry, Rambam Medical Center
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: entacapon.schiz.CTIL
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2005-09

CONDITIONS: Schizophrenia
Keywords: schizophrenia; negative symptoms; entacapone
MeSH Terms: conditions — Schizophrenia | interventions — entacapone

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Entacapone — Entacapone 600mg BID

SUMMARY:
This study is testing the hypothesis that Entacapone added to ongoing antipsychotic treatment can be beneficial in schizophrenic patients with negative symptoms.

ELIGIBILITY:
Inclusion Criteria:

* predominantly negative symptoms
* stable on ongoing antipsychotic treatment

Exclusion Criteria:

* acute psychotic exacerbation
* suicidal ideation
* uncontrolled systemic disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Improvement in specific rating scales during the study and after completion, compared to baseline. | Baseline and once a month untill end of study

SECONDARY OUTCOMES:
Change in PANSS score. | Before and after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ehud Klein, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam medical center, Haifa, Israel